CLINICAL TRIAL: NCT04207606
Title: Follow-up of Pain Intensity Post Epidural Steroid Injection
Brief Title: Post Epidural Steroid Injection Follow-up
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Byron Schneider, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 11192019110246
Record Dates: First submitted 2019-12-10; First posted 2019-12-23 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Lumbago; Lumbar Spinal Stenosis; Lumbar Disc Herniation
Keywords: epidural steroid; lumbar back pain; Pharmacokinetics; Timeline; Natural History
MeSH Terms: conditions — Low Back Pain; Spinal Stenosis; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Epidural Steroid Injection Patients: Patients who are to receive an epidural steroid injection as an outpatient.
  Interventions: Behavioral: Post Epidural Steroid Injection Follow-up

INTERVENTIONS:
Behavioral: Post Epidural Steroid Injection Follow-up — All enrolled patients will undergo epidural steroid injection with fluoroscopy per the Spine Intervention Society guidelines as part of their normal care. Patients will then be contacted for survey responses every 3 days for a maximum of 23 days, to assess pain intensity and change.

SUMMARY:
To determine the expected pain response timeline for patients receiving epidural steroid injections, our team plans to assess patient pain severity and degree of pain relief every 3 days for 23 days.

DETAILED DESCRIPTION:
Patients who are already planning to receive an epidural steroid injection from their physiatrist will be approached by study members on the day of their injection. If enrolled, the patients will be contacted every 3 days for 23 days to determine the severity of pain and degree of pain relief from the injection.

ELIGIBILITY:
Inclusion Criteria:

* Any patient schedule for an epidural steroid injection (ESI) at Stallworth Rehabilitation Hospital through the department of Physical Medicine & Rehabilitation.
* The epidural steroid injection will be performed as part of standard clinical care, this study only aims to describe the clinical response to the procedure.

Exclusion Criteria:

* ESI has been performed within the last 6 months
* Steroid injection elsewhere in body within last 8 weeks
* Oral or intramuscular steroids within last 8 weeks
* Unwilling or unable to provide informed consent
* Unable to comply with required follow up
* Please note that it is assumed that a patient scheduled for an epidural steroid injection clinically is assumed to not have any contraindications to the injection itself such as active systemic infection or pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with low back pain who are to undergo Epidural Steroid Injection for pain relief.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale (NPRS) | post-procedure day 1 (+1 day)
  The NPRS measures pain intensity. Range 0 to 10, with 0 representing "no pain" and 10 representing the worst possible pain. This metric outcome will be the numerical difference between the pre-procedure NPRS score and the NPRS score as measured on post-procedure day 1 (+ 1 day)
Change in Numeric Pain Rating Scale (NPRS) | post-procedure day 4 (+/- 1 day)
  The NPRS measures pain intensity. Range 0 to 10, with 0 representing "no pain" and 10 representing the worst possible pain. This metric outcome will be the numerical difference between the pre-procedure NPRS score and the NPRS score as measured on post-procedure day 4 (+/- 1 day)
Change in Numeric Pain Rating Scale (NPRS) | post-procedure day 7 (+/- 1 day)
  The NPRS measures pain intensity. Range 0 to 10, with 0 representing "no pain" and 10 representing the worst possible pain. This metric outcome will be the numerical difference between the pre-procedure NPRS score and the NPRS score as measured on post-procedure day 7 (+/- 1 day)
Change in Numeric Pain Rating Scale (NPRS) | post-procedure day 10 (+/- 1 day)
  The NPRS measures pain intensity. Range 0 to 10, with 0 representing "no pain" and 10 representing the worst possible pain. This metric outcome will be the numerical difference between the pre-procedure NPRS score and the NPRS score as measured on post-procedure day 10 (+/- 1 day)
Change in Numeric Pain Rating Scale (NPRS) | post-procedure day 13 (+/- 1 day)
  The NPRS measures pain intensity. Range 0 to 10, with 0 representing "no pain" and 10 representing the worst possible pain. This metric outcome will be the numerical difference between the pre-procedure NPRS score and the NPRS score as measured on post-procedure day 13 (+/- 1 day)
Change in Numeric Pain Rating Scale (NPRS) | post-procedure day 16 (+/- 1 day)
  The NPRS measures pain intensity. Range 0 to 10, with 0 representing "no pain" and 10 representing the worst possible pain. This metric outcome will be the numerical difference between the pre-procedure NPRS score and the NPRS score as measured on post-procedure day 16 (+/- 1 day)
Change in Numeric Pain Rating Scale (NPRS) | post-procedure day 19 (+/- 1 day)
  The NPRS measures pain intensity. Range 0 to 10, with 0 representing "no pain" and 10 representing the worst possible pain. This metric outcome will be the numerical difference between the pre-procedure NPRS score and the NPRS score as measured on post-procedure day 19 (+/- 1 day)
Change in Numeric Pain Rating Scale (NPRS) | post-procedure day 22 (+/- 1 day)
  The NPRS measures pain intensity. Range 0 to 10, with 0 representing "no pain" and 10 representing the worst possible pain. This metric outcome will be the numerical difference between the pre-procedure NPRS score and the NPRS score as measured on post-procedure day 22 (+/- 1 day)

SECONDARY OUTCOMES:
Global Rating of Change | Every 3 days for up to 23 days
  Measures reduction in pain intensity. Range: 0 to 100%, with 0% representing no change in pain and 100% representing complete relief of index pain.

CONTACTS AND LOCATIONS:
Overall Officials: Byron J Schneider, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Stallworth Rehabilitation Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No